CLINICAL TRIAL: NCT02371434
Title: The ONE Study: A Unified Approach to Evaluating Cellular Immunotherapy in Solid Organ Transplantation - nTregs Trial
Brief Title: The ONE Study nTreg Trial (ONEnTreg13)
Acronym: ONEnTreg13
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Prof. Dr. Petra Reinke (Other)
Responsible Party: Sponsor-Investigator, Prof. Dr. Petra Reinke, Professor of Nephrology, Charite University, Berlin, Germany
Organization: Charite University, Berlin, Germany (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ONEnTreg13
Record Dates: First submitted 2015-02-18; First posted 2015-02-25 (Estimated); Last update posted 2020-02-05 (Actual); Status verified 2020-02

CONDITIONS: Immunosuppressive Treatment of Living-donor Renal Transplantation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment arm (Experimental): Patients in ONEnTreg13 will be treated with four immunosuppressive agents, all of which are classified as an Investigational Medicinal Products (IMPs):
  * nTregs
  * Prednisolone
  * MMF
  * Tacrolimus
  Interventions: Biological: autologous CD4+CD25+FoxP3+ natural regulat. T cells (nTregs)

INTERVENTIONS:
Biological: autologous CD4+CD25+FoxP3+ natural regulat. T cells (nTregs) — autologous CD4+CD25+FoxP3+ natural regulatory T cells (nTregs). nTregs will be infused at escalating doses of 0.5 x 10^6, 1 x 10^6, and 2.5-3 x 10^6 cells/kg body weight in cohorts of three patients each.

SUMMARY:
The aim of this trial is to collect evidence of the safety of administering autologous CD4+CD25+FoxP3+ natural regulatory T cells (nTregs) to living-donor renal transplant recipients. In addition, the study will determine whether post-transplant nTregs infusion allows a tapering of conventional maintenance immunosuppression within 60 weeks after transplantation.

DETAILED DESCRIPTION:
The ONE Study aims to explore the feasibility, safety and efficacy of regulatory cell therapies as adjunct immunosuppressive treatments in the context of living-donor renal transplantation.The clinical trial presented here (ONEnTreg13) will test autologous, polyclonally expanded CD4+CD25+FoxP3+ nTregs as a somatic cell-based medicinal product.

The objective of this study is to determine whether administration of nTregs to recipients of living-donor kidney transplants is safe and able to polarize the immunological response of the recipient away from graft rejection and towards graft acceptance, allowing a reduction in the doses of pharmacological maintenance immunosuppression.

ELIGIBILITY:
Inclusion Criteria for organ recipients:

* Chronic renal insufficiency with a GFR < 15 ml/min, accepted by the organ transplantation conference, registered by ET (Euro Transplant) and having a positive vote from the living donor ethic commission (Lebendspendekommission) at the Berlin Medical Association.
* Willing and able to participate in The ONE Study IM and HEC Subprojects.
* Signed and dated written informed consent. For patients unable to read and/or write, oral informed consent observed by an independent witness is acceptable if the patient has fully understood oral information given by the Investigator. The witness should sign the consent form on behalf of the patient.

Exclusion Criteria for organ recipients:

* Patient has previously received any tissue or organ transplant other than the planned kidney graft.
* Known contraindication to protocol-specified treatments / medications.
* Genetically identical to the prospective organ donor at the HLA loci, the so called "full house match" (0-0-0 mismatch).
* Panel-Reactive Antibody (PRA) grade > 40% within last 6 months before transplantation.
* Previous treatment with any desensitization procedure (with or without IVIg).
* Concomitant malignancy or history of malignancy within 5 years before study entry (excluding successfully-treated non-metastatic basal/squamous cell carcinoma of the skin).
* Evidence of significant local or systemic infection.
* CMV-negative recipient receiving a kidney from a CMV-positive donor. EBV-negative recipient receiving a kidney from an EBV-positive donor.
* HIV-positive or suffering chronic viral hepatitis.
* Significant liver disease, defined as persistently elevated AST and/or ALT levels > 2 x ULN.
* Malignant or pre-malignant hematological conditions.
* Any uncontrolled medical condition or concurrent disease that could interfere with the study objectives.
* Any condition which, according to the Investigator, would place the subject at undue risk.
* Ongoing treatment with systemic immunosuppressive drugs at study entry.
* Participation in another clinical trial during the study or within 28 days prior to planned study entry.
* Female patients of childbearing potential with a positive pregnancy test at enrolment.
* Female patients who are breast-feeding.
* All female patients of childbearing potential unless the patient is willing to maintain a highly effective method of birth control for the duration of the study.
* Psychological, familial, sociological or geographical factors potentially hampering compliance with the study protocol and follow-up visit schedule.
* Any form of drug or alcohol abuse, psychiatric disorder, or other condition that, in the opinion of the Investigator, may invalidate communication with the Investigator and/or designated study personnel.
* Patients unable to freely give their informed consent (e.g. patients under legal guardianship).
* Patients who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities
* Known allergy/hypersensitivity to any component of the study product.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2015-02; Primary Completion 2017-11-01 (Actual); Study Completion 2017-11-01 (Actual)

PRIMARY OUTCOMES:
Incidence of biopsy-confirmed acute rejection (BCAR) within 60 weeks of organ transplantation | 60 weeks
Incidence of infectious complications associated with cell administration. | 60 weeks
Incidence of embolic pulmonary complications and other embolic events. | 60 weeks
Incidence of immune responses resulting in anaphylactic reactions, cardiovascular compromise or other acute organ failure. | 60 weeks
Biochemical disturbances associated with the cell infusion. | 60 weeks
Over-suppression of the immune system assessed by the incidence of opportunistic infections, especially, CMV, EBV and polyoma virus. | 60 weeks
Over-suppression of the immune system assessed by the incidence of neoplasia. | 60 weeks

SECONDARY OUTCOMES:
Prevention of acute rejection will be secondarily assessed by measuring | 60 weeks
  i) time to first acute rejection episode ii) severity of acute rejection episodes based on response to treatment and histological scoring iii) the level of total immunosuppression drugs at the final trial visit.
Incidence of patients treated for subclinical acute rejection on the basis of histopathological findings | 60 weeks
Prevention of chronic graft dysfunction (chronic rejection or IF/TA) will be assessed by clinical (impairment of GFR) and histopathological (Banff staging) measures. | 60 weeks
Incidence of post-transplant dialysis, inclusion on the transplant waiting list or retransplantation following graft loss through rejection (acute or chronic). | 60 weeks
Avoidance of drug-related complications by immunosuppressant reduction will be assessed by the incidence of reported adverse drug reactions. | 60 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Charité University Medicine, Dept. of Nephrology and Internal Intensive Care, Berlin, Germany

REFERENCES:
- [Derived] Roemhild A, Otto NM, Moll G, Abou-El-Enein M, Kaiser D, Bold G, Schachtner T, Choi M, Oellinger R, Landwehr-Kenzel S, Juerchott K, Sawitzki B, Giesler C, Sefrin A, Beier C, Wagner DL, Schlickeiser S, Streitz M, Schmueck-Henneresse M, Amini L, Stervbo U, Babel N, Volk HD, Reinke P. Regulatory T cells for minimising immune suppression in kidney transplantation: phase I/IIa clinical trial. BMJ. 2020 Oct 21;371:m3734. doi: 10.1136/bmj.m3734. PMID 33087345
- [Derived] Sawitzki B, Harden PN, Reinke P, Moreau A, Hutchinson JA, Game DS, Tang Q, Guinan EC, Battaglia M, Burlingham WJ, Roberts ISD, Streitz M, Josien R, Boger CA, Scotta C, Markmann JF, Hester JL, Juerchott K, Braudeau C, James B, Contreras-Ruiz L, van der Net JB, Bergler T, Caldara R, Petchey W, Edinger M, Dupas N, Kapinsky M, Mutzbauer I, Otto NM, Ollinger R, Hernandez-Fuentes MP, Issa F, Ahrens N, Meyenberg C, Karitzky S, Kunzendorf U, Knechtle SJ, Grinyo J, Morris PJ, Brent L, Bushell A, Turka LA, Bluestone JA, Lechler RI, Schlitt HJ, Cuturi MC, Schlickeiser S, Friend PJ, Miloud T, Scheffold A, Secchi A, Crisalli K, Kang SM, Hilton R, Banas B, Blancho G, Volk HD, Lombardi G, Wood KJ, Geissler EK. Regulatory cell therapy in kidney transplantation (The ONE Study): a harmonised design and analysis of seven non-randomised, single-arm, phase 1/2A trials. Lancet. 2020 May 23;395(10237):1627-1639. doi: 10.1016/S0140-6736(20)30167-7. PMID 32446407